CLINICAL TRIAL: NCT02797535
Title: GI Fluids Collection for an Ex-Vivo Development of Ingestible Capsule Devices With Real Time Biosensors
Acronym: CLARINET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COVGIBD0533
Record Dates: First submitted 2016-04-25; First posted 2016-06-13 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Chronic Inflammatory Small Bowel Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GI fluids samples collection (Other): GI fluids samples will be collected from: (i) fluids suctioned during standard endoscopy procedures / pouchoscopy, (ii) from ileostomy/colostomy bags removed for bag replacement and (iii) from stool samples collected by patients after pouch surgery.
  Interventions: Procedure: Endoscopy procedures

INTERVENTIONS:
Procedure: Endoscopy procedures — GI fluids samples will be collected from: (i) fluids suctioned during standard endoscopy procedures / pouchoscopy, (ii) from ileostomy/colostomy bags removed for bag replacement and (iii) from stool samples collected by patients after pouch surgery.

SUMMARY:
Up to 500 subjects undergoing standard endoscopy / pouchoscopy, or having ileostomy or colostomy bags or having an ileal pouch and who meet the eligibility criteria will be enrolled to this study during up to three years at up to 4 clinical sites. GI fluids samples will be collected from: (i) fluids suctioned during standard endoscopy procedures / pouchoscopy, (ii) from ileostomy/colostomy bags removed for bag replacement and (iii) from stool samples collected by patients after pouch surgery.

DETAILED DESCRIPTION:
Up to 500 subjects undergoing standard endoscopy / pouchoscopy, or having ileostomy or colostomy bags or having an ileal pouch and who meet the eligibility criteria will be enrolled to this study during up to three years at up to 4 clinical sites. GI fluids samples will be collected from: (i) fluids suctioned during standard endoscopy procedures / pouchoscopy, (ii) from ileostomy/colostomy bags removed for bag replacement and (iii) from stool samples collected by patients after pouchsurgery.

The samples will be collected into sealed plastic containers, clearly labeled with "Biohazard" stickers and patient's code and be kept on ice for up to 30min and then freezed in -20deg to -80deg.

Characterization and quanification of small molecules- and protein biomarkers of GI diseases such as IBD will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ages 18-75 years
* Subjects referred to endoscopic procedures gastroscopy, esophagogastroduodenoscopy (EGD), colonoscopy, single balloon or double balloon enteroscopy Or Subjects having ileostomy or colostomy bags Or Subjects having an ileal pouch
* Subjects agree to sign consent form

Exclusion Criteria:

* Patients has any medical condition that requires special handling of body fluids beyond routine infection control measures (i.e. standard surgical gloves)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Characterization and quantification of small molecules- and protein biomarkers of GI diseases will be performed. Examples of such biomarkers include - calprotectin, lactoferrin, albumin, hemoglobin, CEA, CA19-9, CA 72-4, LYVE-1, REG1A, TFF1 and ammonia. | 3 years
  The concentration of the biomarkers in the collected fluids from different parts of the GI will be determined by quantitative assays - such as ELISA or lateral flow immunoassay or mass spectrometry. Concentration will be determined in mg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Rami Eliakim, Prof., Principal Investigator — Sheba Medical Center
Locations (2):
- Israel (2):
  - Sheba Medical Center, Ramat Gan
  - The Tel-Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No